CLINICAL TRIAL: NCT05217056
Title: Associations Between General Movements Assessments and Cognitive Development in a Cohort of High Risk of Infants: One Year Follow Up
Brief Title: Associations Between General Movements Assessments and Cognitive Development
Acronym: GMs
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Hatice Adiguzel, Assistant Proffessor, Kahramanmaras Sutcu Imam University
Other Study IDs: KSU2
Record Dates: First submitted 2022-01-05; First posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Cerebral Palsy; Infant Development; Cognitive Dysfunction; Cognitive Developmental Delay; Cognitive Impairment, Mild; Infant, Small for Gestational Age; Infant, Premature, Diseases; Infant Asphyxia; Infant, Very Low Birth Weight
Keywords: General Movements(GMs); Cognitive Development; BAYLEY-III Infant and Toddler Development Assessment; High Risk of Infants
MeSH Terms: conditions — Cerebral Palsy; Cognitive Dysfunction; Infant, Premature, Diseases | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/Measurement: All of the infants with high risk of cerebral palsy
  Interventions: Other: measurements

INTERVENTIONS:
Other: measurements — All of the infants with high risk of cerebral palsy will be assessed from birth to 12 months age with the assessments of Prechtl's General movements (GMs) until 20 weeks of age. Also BAYLEY-III Infant and Toddler Development Assessment Scale (BAYLEY-III) will be performed at the 3rd, 6th, and 12th months for the cognitive development.

SUMMARY:
High risk infant is defined as infant with a negative history of environmental and biological factors, which can lead to neuromotor development problems. It is a heterogeneous group of premature infants born under thirty-seven weeks of age, with infants with low birth weight, term or developmental retardation for various reasons. Therefore, preterm infants with low birth weight can survive with a neurological sequelae such as cerebral palsy (CP), epilepsy, hearing and vision loss, mental retardation, speech and speech problems, and learning difficulties. The clinical diagnosis of CP and learning diffuculties which can be observed in high-risk infants, is based on the combination of some neurological and clinical signs.

DETAILED DESCRIPTION:
High-risk of infant follow-up programs provide guidance for the treatment of neurodevelopmental delays and deterioration in terms of early development. Three methods with the best predictable validity that can determine CP before the adjusted age of 5-month is Magnetic Resonance Imaging (MRI), Prechtl's Assessment of General Movements (GMs), Hammersmith Infant Neurological Evaluation. In recent years, the diagnosis of high-risk of CP can be detected at 3 months with predictive validity and reliability by evaluating the quality of GMs. GMs are now considered the gold standard for early detection of CP because of its high sensitivity and specificity than MRI, cranial US and neurological evaluations. It was also found that cognitive or language skills may be inadequate in school age in patients with inadequate movement character and in the same postural patterns according to age, although GMs are normal. So new clinical care guidelines and new intervention research for infants with CP and learning diffuculties under the age of 1, needs to be been shown. There a few studies about early detection of learning diffuculties like autism spectrum disorders between GMs and cognitive development tests. So this study aimed to reveal the association between GMs and cogtinive development with a cohort of high risk of infants with one year floow up.

ELIGIBILITY:
Inclusion Criteria:

* Having periventricular hemorrhage, ICH stages 2, 3, 4, cystic PVL, stage 3 HIE, kernicterus, perinatal asphyxia, chronic lung disease, RDS, BPD, long-term oxygen (7 days), >24 hours mechanical ventilator (MV) support, 5th minute Apgar Score <3, neonatal sepsis, necrotizing enterocolitis (NEC), retinopathy of prematurity (ROP), gestation age <32 weeks, and prematurity due to preterm/multiple births<1500 gr.

Exclusion Criteria:

* Infants with congenital malformation (Spina Bifida, Congenital Muscular Torticollis, Arthrogriposis Multiplex Congenita etc.)
* Infants diagnosed with metabolic and genetic diseases (Down Syndrome,Spinal Muscular Atrophy, Duchenne Muscular Dystrophy etc.)
* Infants still intubated and mechanical ventilator dependent at postterm 3 months

Ages: 25 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: high risk of infanst for cerebral palsy
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Prechtl's General movements (GMs) assessments1 | Measurement at preterm age (birth to 40weeks)
  General movements (GMs) are the spontaneous movement repertoire present from early foetal life until 20 weeks post-term. From birth to 8 post-term weeks, they have a "writhing" character. They will be scored as cs-pr-n-ch. N show normal movement patterns.
Prechtl's General movements (GMs) assessments2 | Measurement between the term age to 9th weeks
  General movements (GMs) are the spontaneous movement repertoire present from early foetal life until 20 weeks post-term. From birth to 8 post-term weeks, they have a "writhing" character. They will be scored as cs-pr-n-ch. N show normal movement patterns.
Prechtl's General movements (GMs) assessments3 | Measurement at fidgety periods of life (between 10th weeks to 20th weeks)
  General movements (GMs) are the spontaneous movement repertoire present from early foetal life until 20 weeks post-term. From birth to 8 post-term weeks, they have a "writhing" character and then till about 20 weeks a "fidgety" character. Two specific abnormal movement patterns reliably predict CP in fidgety term: F (-): the absence of the fidgety character from 8-20 post-term weeks. Fidgety movements (FMs) are classified as (a) normal (F+), (b) absent (AF), when normal FMs are never observed and (c) abnormal (F-).
The Bayley Scales of Infant and Toddler Development, Third Edition (BSID-III) | Change from the baseline of the BAYLEY-III score at 3, 6,12th month of infants
  The BSID-III is a neurocognitive assessment used to evaluate infants from 0-42 months and to monitor their development with 5 domains: cognitive, language (receptive and expressive communication), motor (fine and gross motor), social-emotional, and adaptive functions (17). The first three domains will be assessed. To allow comparison of results from the 5 domains, a composite score will be calculated for each domain (mean, 100±15). A composite score below -2 standard deviation (SD) (<70) will be considered a severe delay for all domains.

SECONDARY OUTCOMES:
demographic information1 | first day of birth
  birth age of the infants will be recorded in weeks
demographic information2 | first day of birth
  birth weight of the infants will be recorded in kilograms

CONTACTS AND LOCATIONS:
Overall Officials: hatice adıgüzel, PhD, Principal Investigator — Kahramanmaras Sutcu Imam University; Bulent Elbasan, Proffessor, Study Director — Gazi University
Locations (1):
- Hatice Adıgüzel, Kahramanmaraş, Dulkadiroglu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No